CLINICAL TRIAL: NCT04786990
Title: A Phase IV, Open-Label, Flexible-Dose Safety Trial Evaluating SPN-812 Administered With Psychostimulants in Children and Adolescents (6 to 17 Years of Age) With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Open-Label Study of SPN-812 Administered With Psychostimulants in Children and Adolescents With ADHD
Acronym: ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812P412
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Treatment (Experimental): Subjects 6-11 years of age: 100 to 400mg SPN-812 (100 mg oral capsule)
  Subjects 12-17 years of age: 100 to 600mg SPN-812 (100 mg, 200 mg oral capsule)
  Interventions: Drug: SPN-812

INTERVENTIONS:
Drug: SPN-812 — Viloxazine extended-release capsule

SUMMARY:
This open label, flexible-dose study evaluating the safety and efficacy of SPN-812 administered with psychostimulants in children and adolescents (6 to 17 years of age) with Attention-Deficit/Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This is an open-label, multicenter, flexible-dose, safety study of SPN-812 in pediatric patients (6-17 years of age) diagnosed with ADHD, when administered with a FDA-approved medication (psychostimulant) in the treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in pediatric subjects. Participants will be screened for eligibility for up to 4 weeks, and he/she will continue to take their prescribed psychostimulant ADHD medication during that time. Following the screening period, eligible subjects will receive SPN-812 with their current psychostimulant treatment for ADHD for 8 weeks. For the first 4 weeks of treatment subjects will take SPN-812 dose in the morning (AM dosing), and for the last 4 weeks of treatment, subjects will take SPN-812 dose in the evening (PM dosing). The total duration of the study between the screening visit and the end of the treatment period/end of study (EOS) visit is up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, 6 to ≤17 years and 9 months of age at screening.
2. Parent(s)/legal guardian(s) is able to read and understand the Informed Consent Form (ICF).
3. Written informed consent obtained by parent(s)/legal guardian(s) and informed assent obtained from the subject, if applicable.
4. Subject and parent(s)/legal guardian(s) are willing and able to comply with all of the procedures and requirements defined in the protocol, including parents(s)/legal guardian(s) oversight of morning and evening dosing of the SPN-812 and recording a daily medication/dosing diary for psychostimulant and/or SPN-812 during the study.
5. Has lived with the same parent(s)/legal guardian(s) at same residence for at least the last 6 months prior to screening.
6. Has a primary diagnosis of ADHD (inattentive, hyperactive, or combined presentation) confirmed with the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) at screening.
7. Is currently on a single, stable psychostimulant regimen (see Inclusion Criterion 8 for definition) for treatment of ADHD with a partial, but inadequate efficacy response to at least 2 weeks of treatment with a psychostimulant (methylphenidate or amphetamine) prior to screening. An inadequate response is defined as an investigator-rated ADHD-RS-5 Total score ≥24 and a CGI-S score ≥3 (mildly ill or worse) at Screening and Baseline. Subjects taking additional medication for ADHD (e.g., nonstimulant) are excluded.
8. Is currently and expecting to continue and remain on a stable psychostimulant regimen throughout the study. A stable stimulant regimen is defined as taking dose at least 5 days per week (morning), no significant change in dose or dosing frequency at least 2 weeks prior to baseline (Visit 2), and the investigator believes the subject's psychostimulant dose is optimized.
9. Is functioning at an age-appropriate level intellectually, as judged by the Investigator.
10. Is a child (6-11 years of age) with a body weight of at least 20 kg at screening or is an adolescent (12-17 years of age) with a body weight of at least 35 kg at screening.
11. Has a resting (sitting) blood pressure (BP) and resting pulse rate measurement within the 95th percentile for age, sex, and height.
12. Is considered medically healthy by the Investigator via assessment of physical examination, medical and psychiatric histories, clinical laboratory tests, vital signs, and electrocardiogram (ECG).
13. Females of childbearing potential (FOCP) must be either sexually inactive (abstinent) or, if sexually active, must agree to use/practice one of the following acceptable, highly effective contraceptive methods beginning/during the screening period prior to the first dose of SM and throughout the study:

    1. Simultaneous use of male condom and intra-uterine contraceptive device placed during screening period prior to first dose of SM
    2. Surgically sterile male partner (e.g., vasectomized partner is sole partner)
    3. Barrier method: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
    4. Established use of oral, injected, or implanted hormonal methods of contraception

    With approval by the Investigator, subjects' parents or legal guardians may select abstinence as a form of birth control if deemed more appropriate. For the purposes of this study, all females are considered to be of childbearing potential unless they are confirmed by the Investigator to be premenarchal, biologically sterile, or surgically sterile (e.g., hysterectomy with bilateral oophorectomy, tubal ligation).
14. Adolescent males, if sexually active, must:

    1. Use 2 methods of contraception in combination if his female partner is of childbearing potential; this combination of contraceptive methods must be used from the Baseline Visit to ≥ 1 month after the last dose of SM, or
    2. Have been surgically sterilized prior to the Screening Visit.

Exclusion Criteria:

1. Is currently participating in another clinical trial or has participated in a clinical trial within 60 days prior to screening.
2. Is a member of the study personnel or of their immediate families, or is a subordinate (or immediate family member of a subordinate) to any of the study personnel.
3. Is a female subject who is pregnant, lactating and/or sexually active and not agreeing to use one of the acceptable contraceptive methods throughout the study.
4. Has history of severe drug allergy or hypersensitivity, or known hypersensitivity, to the study medication (SPN-812).
5. Has history of moderate or severe head trauma or other neurological disorder or systemic medical disease that, in the Investigator's opinion, is likely to affect central nervous system functioning. This would include subjects with:

   1. a current diagnosis of a major neurological disorder;
   2. seizures, seizure disorder or seizure-like events;
   3. history of seizure disorder within the immediate family (siblings, parents); or
   4. encephalopathy

   Note: Febrile seizures are not exclusionary and will be assessed on a case-by-case basis. If for any reason the subject received medication for a febrile seizure or has a history of complex febrile seizures, this will be exclusionary.
6. Has current diagnosis or history of major psychiatric disorders or intellectual disabilities other than ADHD per DSM-5 criteria (including schizophrenia, schizoaffective disorder, bipolar disorder, borderline personality disorder, antisocial personality disorder, narcissistic personality disorder, post-traumatic stress disorder, obsessive-compulsive disorder, severe oppositional defiant disorder (ODD), conduct disorder, and disruptive mood dysregulation disorder, and autism spectrum disorders). The following is not exclusionary:

   1. a history of mild social anxiety disorder or generalized anxiety disorder according to DSM-5 criteria;
   2. a history of mild to moderate ODD according to DSM-5 criteria;
   3. a history of Major Depressive Disorder, if he/she has not experienced a major depressive disorder episode or required psychiatric counselling; or pharmacotherapy within the 6 months prior to screening
7. Has a known history of physical, sexual, or emotional abuse in the last year prior to screening.
8. Has any other disorder for which its treatment takes priority over treatment of ADHD or is likely to interfere with study treatment, impair treatment compliance, or interfere with interpretation of study results.
9. Has a current diagnosis of drug abuse or dependence disorder within the 12 months prior to screening, has a history of drug abuse or dependence disorder or has an immediate family member living at study participant's' home who has current diagnosis drug abuse or dependence disorder (per DSM-5 criteria).
10. Evidence of suicidality (defined as either active suicidal plan/intent or active suicidal thoughts, or more than one lifetime suicide attempt) within the six months before Screening or at Screening.
11. Has positive findings on C-SSRS for suicidal ideation or behaviors at screening. Has attempted suicide within the 6 months prior to screening, or is at significant risk of suicide, either in the opinion of the Investigator or defined as a "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behavior on the C-SSRS within the 6 months prior to screening.
12. Is currently using, or has a positive result on the urine drug screening for, drugs of abuse (alcohol, amphetamine, barbiturates, benzodiazepines, cannabis [THC], cocaine, cotinine, methadone, methamphetamine [including ecstasy], methylphenidate, phencyclidine, propoxyphene, and opiates) with the exception of the psychostimulant prescribed for the treatment of ADHD.
13. Is unable to discontinue all prohibited medication at least 7 days prior to baseline.
14. Has body mass index (BMI) greater than 95th percentile for her/his appropriate age and gender (per CDC's gender specific "BMI-for-age percentiles" charts).
15. Has a current diagnosis of significant systemic disease.
16. Has uncontrolled thyroid disorder defined as thyroid stimulating hormone ≤ 0.8 x the lower limit of normal or ≥ 1.25 x the upper limit of normal for the reference laboratory range.
17. Has resting (sitting) blood pressure and pulse rate greater than the 95th percentile for age and gender.
18. Has a known personal history, or presence, of structural cardiac abnormalities, cardiovascular or cerebrovascular disease, serious heart rhythm abnormalities, syncope, tachycardia, cardiac conduction problems (e.g., clinically significant heart block or QT interval prolongation: QTc >0.44 seconds), exercise-related cardiac events including syncope and pre-syncope, or clinically significant bradycardia.
19. Has any clinically significant abnormal clinical laboratory test, urine test, electrocardiogram (ECG) result, vital signs or physical examination finding at screening that, in the opinion of the Investigator, would interfere with the safety of the subject
20. Has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments.
21. Has or has had one or more medical conditions considered clinically significant/relevant by the Investigator in the context of the study (e.g., cardiovascular disease, congestive heart failure, cardiac hypertrophy, arrhythmia, bradycardia [pulse < 70 bpm (6-11 years), pulse < 60 bpm (12-17 years)], tachycardia [pulse > 120 bpm (6-11 years); pulse > 100 bpm (12-17 years)], respiratory disease, hepatic impairment or renal insufficiency, metabolic disorder, endocrine disorder, gastrointestinal disorder, hematological disorder, infectious disorder, any clinically significant immunological condition, dermatological disorder.
22. Has any disease or medication that could, in the Investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with study conduct or interpretation of results.
23. Lost or donated more than 450 mL of blood during the 30 days prior to screening.
24. Use of any investigational drug or prohibited concomitant medications including known CYP1A2 substrates (e.g., theophylline, melatonin) within 28 days or 5 half-lives prior to Baseline Visit (Day 1) (whichever is longer) or anticipated for the duration of the study.
25. History of unexplained loss of consciousness, unexplained syncope, unexplained irregular heartbeats or palpitations or near drowning with hospital admission.
26. Has an allergy to applesauce and cannot swallow capsules whole.
27. In the Investigator's opinion, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, MBA, Study Director — Chief Medical Officer
Locations (17):
- United States (16):
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - NRC Research Institute, Orange, California
  - Miami Clinical Research, Miami, Florida
  - APG Research, LLC, Orlando, Florida
  - Elite Clinical Trials, Blackfoot, Idaho
  - Elite Clinical Trials, Rexburg, Idaho
  - Qualmedica Research, LLC, Evansville, Indiana
  - Psychiatric Associates Purehealth Medical Center, Overland Park, Kansas
  - Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Gadolin Research, LLC, Beaumont, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Barbara Diaz Hernandez MD Research, INC., San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Treatment: SPN-812 (viloxazine extended-release capsules)
  Subjects 6-11 years of age: 100 to 400mg SPN-812 (100 mg oral capsule)
  Subjects 12-17 years of age: 100 to 600mg SPN-812 (100 mg, 200 mg oral capsule)
Period: Overall Study
Arm/Group | Open-Label Treatment
Started (Number of subjects "Started" is based on the Safety Population (defined as subjects who signed an Informed Consent and took at least one dose of SPN-812).) | 56
Completed | 48
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Noncompliance | 1
Not completed — Unable to complete site visits | 1
Not completed — Withdrawal by Parent/Guardian | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (2.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 45
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 56
Investigator-rated Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (IR-ADHD-RS-5) [Mean (Standard Deviation); unit: units on a scale] — The Investigator-rated Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (IR-ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Each item was rated by a trained investigator on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). Sum of all 18 items yields the raw Total score (range: 0-54; the higher the score, the more severe the ADHD symptoms).
  units on a scale | 37.2 (8.35)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events During 8 Weeks of Adjunct SPN-812 Treatment
Description: The percent of subjects who took at least one dose of SPN-812 and reported at least one adverse event during 8 weeks of adjunct SPN-812 Treatment. The percent is calculated by dividing "the number of subjects who reported at least one Adverse Event (n)" by "the number of subjects in the Safety Population (N)" and then multiplying the product by 100. The higher the percent, the higher the incidence.
Time Frame: Weeks 1-8
Population: Safety Population, defined as subjects who signed Informed Consent and took at least one dose of SPN-812.
Measure: Number; unit: percent of subjects
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
percent of subjects | 55.4

2. Secondary Outcome: Incidence of Adverse Events During Adjunctive SPN-812 Treatment During Weeks 1-4 (SPN-812 Dosed in Morning Hours [AM Dosing]) and During Weeks 5-8 (SPN-812 Dosed in Evening Hours [PM Dosing])
Description: The percent of subjects who reported at least one adverse event during adjunctive SPN-812 Treatment during Weeks 1-4 (SPN-812 dosed in morning hours [AM Dosing]) and during Weeks 5-8 (SPN-812 dosed in evening hours [PM Dosing]). The percent is calculated by dividing "the number of subjects who reported at least one Adverse Event (n) during Weeks 1-4 or Weeks 5-8" by "the number of subjects analyzed during Weeks 1-4 or Weeks 5-8" (subjects who took at least once dose of SPN-812 during Weeks 1-4 or Weeks 5-8), respectively and then multiplying the product of each by 100. The higher the percent, the higher the incidence.
Time Frame: Weeks 1-4 and Weeks 5-8
Population: Safety Population, defined as subjects who signed Informed Consent and took at least one dose of SPN-812. The data (percent of subjects who reported at least one adverse event for Weeks 1-4 or Weeks 5-8) is summarized by the number of subjects analyzed (subjects who took at least one dose of SPN-812 during Weeks 1-4 or Weeks 5-8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Number; unit: Percent of subjects
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
Percent of subjects
  Percent of subjects; Weeks 1-4 | 50.0
  Percent of subjects; Weeks 5-8: number analyzed (Participants) | 50
  Percent of subjects; Weeks 5-8 | 36.0

3. Secondary Outcome: Change From Baseline in the Investigator-rated Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (IR-ADHD-RS-5) Total Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Each item was rated by a trained investigator on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). The sum of all 18 items yields the raw Total score (range: 0-54; the higher the score, the more severe the ADHD symptoms). Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data at each Week/Visit is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid Investigator-rated ADHD Rating Scale, 5th Edition [IR-ADHD-RS-5] assessment at baseline [pre-dosing] and at Week 4 or Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Open-Label Treatment: SPN-812 (viloxazine extended-release capsules)
  Subjects 6-11 years of age: 100 to 400 mg SPN-812 (100 mg oral capsule)
  Subjects 12-17 years of age: 100 to 600 mg SPN-812 (100 mg, 200 mg oral capsule)
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline | 37.2 (8.35)
  Change from Baseline score; Week 4: number analyzed (Participants) | 54
  Change from Baseline score; Week 4 | -13.5 (9.70)
  Change from Baseline score; Week 8: number analyzed (Participants) | 48
  Change from Baseline score; Week 8 | -18.2 (9.99)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — The p-value generated from the statistical test for this efficacy measure is considered nominal. An adjustment for multiplicity was not performed, and as a result, there is no control of Type 1 error in the statistical analysis of these data
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Severity of Illness (CGI-S) Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Clinical Global Impression-Severity of Illness (CGI-S) scale is a single item clinician-rated assessment of the severity of the ADHD symptoms in relation to the clinician's total experience with patients with ADHD. The CGI-S is evaluated by the investigator on a 7-point scale, where 1 = Normal, not at all ill; 2 = Borderline mentally Ill; 3 = Mildly Ill; 4 = Moderately Ill; 5 = Markedly Ill; 6 = Severely Ill; and 7 = Among the most extremely ill patients; the higher the score, the more severe the ADHD symptoms. Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: Safety population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data at each Week/Visit is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid Clinical Global Impression-Severity of Illness Scale [CGI-S] assessment at baseline [pre-dosing] and at Week 4 or Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline | 4.4 (0.56)
  Change from Baseline score; Week 4: number analyzed (Participants) | 54
  Change from Baseline score; Week 4 | -0.9 (0.92)
  Change from Baseline score; Week 8: number analyzed (Participants) | 48
  Change from Baseline score; Week 8 | -1.4 (1.10)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Clinical Global Impression-Improvement (CGI-I) is a single item, clinician-rated assessment of how much the clinician believes the subject's overall symptoms have changed (improved, worsened or no change) relative to subject's baseline state prior to the beginning of treatment. The CGI-I is evaluated by the investigator on a 7-point scale, where 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, and 7 = Very much worse. A CGI-I score <4 represents a better outcome.
Time Frame: Week 4 and Week 8
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data at each Week/Visit is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid Clinical Global Impression-Improvement [CGI-I] assessment at Week 4 or Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Open Label Treatment: SPN-812 (viloxazine extended-release capsules)
  Subjects 6-11 years of age: 100 to 400 mg SPN-812 (100 mg oral capsule)
  Subjects 12-17 years of age: 100 to 600 mg SPN-812 (100 mg, 200 mg oral capsule)
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Week 4: number analyzed (Participants) | 54
  Raw score; Week 4 | 2.8 (0.95)
  Raw score; Week 8: number analyzed (Participants) | 48
  Raw score; Week 8 | 2.3 (0.97)

6. Secondary Outcome: Change From Baseline in the Sleep Disturbance Scale for Children (SDSC) Total Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six Subscale scores are generated: (1) disorders of initiating and maintaining sleep (7 items), (2) sleep breathing disorders (3 items), (3) disorders of arousal (3 items), (4) sleep-wake transition disorders (6 items), (5) disorders of excessive somnolence (5 items), and (6) sleep hyperhidrosis (2 items). The sum of all Subscale scores yields the raw Total score (range: 26 to 130; the higher the score, the more severe sleep disturbance). Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data at each Week/Visit is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid Sleep Disturbance Scale for Children [SDSC] assessment at baseline [pre-dosing] and at Week 4 or at Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 54.4 (17.75)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -8.8 (14.03)
  Change from Baseline score; Week 8: number analyzed (Participants) | 46
  Change from Baseline score; Week 8 | -10.3 (17.39)
Statistical Analysis 1: Comparison: Open Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open Label Treatment; Week 8; Test type: Other; p = 0.0002, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline in the Sleep Disturbance Scale for Children (SDSC) "Disorders of Initiating and Maintaining Sleep (DIMS)" Subscale Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Disorders of Initiating and Maintaining Sleep (DIMS) Subscale (items 1,2,3,4,5,10, and 11). The sum of the 7 items yields the raw Subscale score (range: 7 to 35; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 19.9 (6.38)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -3.2 (4.84)
  Change from Baseline score; Week 8: number analyzed (Participants) | 46
  Change from Baseline score; Week 8 | -4.2 (6.08)
Statistical Analysis 1: Comparison: Open Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open Label Treatment; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided — The p-value generated for the comparison between time points for this efficacy measure is considered nominal. An adjustment for multiplicity was not performed. There is no control of Type 1 error in the statistical analysis of these data

8. Secondary Outcome: Change From Baseline in the Sleep Disorders Scale for Children (SDSC) "Sleep Breathing Disorder (SBD)" Subscale Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Sleep Breathing Disorder (SBD) Subscale (items 13, 14, and 15). The sum of the 3 items yields the raw Subscale score (range: 5 to 15; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 4.2 (2.07)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -0.5 (1.85)
  Change from Baseline score; Week 8: number analyzed (Participants) | 46
  Change from Baseline score; Week 8 | -0.3 (2.06)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p = 0.0685, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p = 0.2575, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

9. Secondary Outcome: Change From Baseline in the Sleep Disturbance Scale for Children (SDSC) "Disorders of Arousal (DA)" Subscale Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Disorders of Arousal (DA) Subscale (items 17, 20, and 21). The sum of the 3 items yields the raw Subscale score (range: 5 to 15; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 3.9 (1.50)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -0.3 (1.17)
  Change from Baseline score; Week 8: number analyzed (Participants) | 46
  Change from Baseline score; Week 8 | -0.2 (1.47)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p = 0.0832, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p = 0.3715, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

10. Secondary Outcome: Change From Baseline in the Sleep Disturbance Scale for Children (SDSC) "Sleep-Wake Transition Disorders (STD)" Subscale Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Sleep-Wake Transition Disorders (STD) Subscale (items 6, 7, 8, 12, 18, and 19). The sum of the 6 items yields the raw Subscale score (range: 6 to 30; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 11.8 (5.13)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -1.8 (4.49)
  Change from Baseline score; Week 8: number analyzed (Participants) | 46
  Change from Baseline score; Week 8 | -2.5 (5.04)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p = 0.0042, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p = 0.0019, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

11. Secondary Outcome: Change From Baseline in the Sleep Disorders Scale for Children (SDSC) "Disorders of Excessive Somnolence (DES)" Subscale Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Disorders of Excessive Somnolence (DES) Subscale (items 22, 23, 24, 25, and 26). The sum of the 5 items yields the raw Subscale score (range: 5 to 25; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 11.0 (4.66)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -2.3 (3.87)
  Change from Baseline score; Week 8: number analyzed (Participants) | 46
  Change from Baseline score; Week 8 | -2.3 (4.87)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p = 0.0025, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

12. Secondary Outcome: Change From Baseline in the Sleep Disorders Scale for Children (SDSC) "Sleep Hyperhidrosis (SH)" Subscale Scores at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Sleep Hyperhidrosis (SH) Subscale (items 9 and 16). The sum of the 2 items yields the raw Subscale score (range: 2 to 10; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 3.7 (2.61)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -0.7 (1.99)
  Change from Baseline score; Week 8: number analyzed (Participants) | 46
  Change from Baseline score; Week 8 | -0.8 (2.03)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p = 0.0161, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p = 0.0122, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

13. Secondary Outcome: Change From Baseline in Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) Total Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) is a validated, 11-item scale for the assessment of ADHD-related morning and evening behaviors impacting at-home functioning in children with ADHD. There are 3 items related to morning behaviors and 8 items related to evening behaviors. The parent/guardian rates each item on a 4-point scale based on their child's behavior during the past week, where 0 = "no difficulty" to 3 = "a lot of difficulty". The sum of all 11 items yields a Total score (range: 0-33); the higher the score, the more severe the impairment/difficulty. Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data at each Week/Visit is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid Weekly Parent Rating of Evening and Morning Behavior-Revised [WPREMB-R] assessment at baseline [pre-dosing] and at Week 4 or at Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 19.6 (6.39)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -5.2 (6.03)
  Change from Baseline score; Week 8: number analyzed (Participants) | 47
  Change from Baseline score; Week 8 | -7.7 (6.87)
Statistical Analysis 1: Comparison: Open Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open Label Treatment; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

14. Secondary Outcome: Change From Baseline in Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) "Morning Behaviors" Subscale Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) is a validated, 11-item scale for the assessment of ADHD-related morning and evening behaviors impacting at-home functioning in children with ADHD. There are 3 items related to morning behaviors and 8 items related to evening behaviors. The parent/guardian rates each item on a 4-point scale based on their child's behavior during the past week, where 0 = "no difficulty" to 3 = "a lot of difficulty". The sum of all 3 items related to morning behaviors yields a WPREMB-R Morning Behaviors Subscale score (range: 0-9); the higher the score, the more severe the impairment/difficulty. Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 5.4 (2.32)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -1.2 (2.18)
  Change from Baseline score; Week 8: number analyzed (Participants) | 47
  Change from Baseline score; Week 8 | -1.6 (2.24)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p = 0.0002, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

15. Secondary Outcome: Change From Baseline in Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) "Evening Behaviors" Subscale Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) is a validated, 11-item scale for the assessment of ADHD-related morning and evening behaviors impacting at-home functioning in children with ADHD. There are 3 items related to morning behaviors and 8 items related to evening behaviors. The parent/guardian rates each item on a 4-point scale based on their child's behavior during the past week, where 0 = "no difficulty" to 3 = "a lot of difficulty". The sum of all 8 items related to evening behaviors yields a WPREMB-R Evening Behaviors Subscale score (range: 0-24); the higher the score, the more severe the impairment/difficulty. Raw score is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 55
  Raw score; Baseline | 14.2 (5.00)
  Change from Baseline score; Week 4: number analyzed (Participants) | 53
  Change from Baseline score; Week 4 | -4.1 (4.44)
  Change from Baseline score; Week 8: number analyzed (Participants) | 47
  Change from Baseline score; Week 8 | -6.1 (5.27)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

16. Secondary Outcome: Change From Baseline in the Investigator-rated Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (IR-ADHD-RS-5) Total Score at Week 4 (AM Dosing) Versus Week 8 (PM Dosing)
Description: The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Each item was rated by a trained investigator on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). The sum of all 18 items yields the raw Total score (range: 0-54; the higher the score, the more severe the ADHD symptoms). Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: Safety population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data is summarized by number of subjects analyzed (n; subjects with a valid Investigator-rated ADHD Rating Scale, 5th Edition [IR-ADHD-RS-5] assessment at baseline [pre-dosing], Week 4, and Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 48
score on a scale | -4.8 (8.90)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.0005, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

17. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Illness (CGI-S) Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Clinical Global Impression-Severity of Illness (CGI-S) scale is a single item clinician-rated assessment of the severity of the ADHD symptoms in relation to the clinician's total experience with patients with ADHD. The CGI-S is evaluated by the investigator on a 7-point scale, where 1 = Normal, not at all ill; 2 = Borderline mentally Ill; 3 = Mildly Ill; 4 = Moderately Ill; 5 = Markedly Ill; 6 = Severely Ill; and 7 = Among the most extremely ill patients; the higher the score, the more severe the ADHD symptoms. Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: Safety population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data is summarized by number of subjects analyzed (n; subjects with a valid Clinical Global Impression-Severity of Illness Scale [CGI-S] assessment at baseline [pre-dosing], Week 4, and Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 48
score on a scale | -0.5 (0.97)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.0005, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

18. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Clinical Global Impression-Improvement (CGI-I) is a single item, clinician-rated assessment of how much the clinician believes the subject's overall symptoms have changed (improved, worsened or no change) relative to subject's baseline state prior to the beginning of treatment. The CGI-I is evaluated by the investigator on a 7-point scale, where 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, and 7 = Very much worse. A mean difference (the Week 8 minus the Week 4 CGI-I score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: Safety population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid Clinical Global Impression-Improvement [CGI-I] assessment at Week 4 and Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 48
score on a scale | -0.5 (0.99)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.0016, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

19. Secondary Outcome: Change From Baseline in Sleep Disturbance Scale for Children (SDSC) Total Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". 6 Subscale scores are generated: 1) disorders of initiating and maintaining sleep, 7 items; 2) sleep breathing disorders, 3 items; 3) disorders of arousal, 3 items; 4) sleep-wake transition disorders, 6 items; 5) disorders of excessive somnolence, 5 items; and 6) sleep hyperhidrosis, 2 items. Sum of all Subscale scores yields a raw Total score (range: 26 to 130; higher score indicates more severe sleep disturbance). Raw score is converted to a change from baseline (CFB) score. A mean difference (Week 8 minus Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data is summarized by number of subjects analyzed (n; subjects with a valid Sleep Disturbance Scale for Children [SDSC] assessment at baseline [pre-dosing], Week 4, and Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 46
score on a scale | -0.2 (9.54)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.8900, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

20. Secondary Outcome: Change From Baseline in Sleep Disorders Scale for Children (SDSC) "Disorders of Initiating and Maintaining Sleep (DIMS)" Subscale Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Disorders of Initiating and Maintaining Sleep (DIMS) Subscale (items 1, 2, 3, 4, 5, 10, and 11). The sum of the 7 items yields the raw Subscale score (range: 7 to 35; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 46
score on a scale | -0.5 (3.57)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.3269, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

21. Secondary Outcome: Change From Baseline in Sleep Disorders Scale for Children (SDSC) "Sleep Breathing Disorder (SBD)" Subscale Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Sleep Breathing Disorder (SBD) Subscale (items 13, 14, and 15). The sum of the 3 items yields the raw Subscale score (range: 5 to 15; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 46
score on a scale | 0.2 (1.55)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.5085, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

22. Secondary Outcome: Change From Baseline in Sleep Disturbance Scale in Children (SDSC) "Disorders of Arousal (DA)" Subscale Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Sleep Disorders Scale for Children (SDSC) is a 26-item, parent-reported measure used to screen for sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Disorders of Arousal (DA) Subscale (items 17, 20, and 21). The sum of the 3 items yields the raw Subscale score (range: 5 to 15; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 46
score on a scale | 0.1 (0.93)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.3484, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

23. Secondary Outcome: Change From Baseline in Sleep Disorders Scale for Children (SDSC) "Sleep-Wake Transition Disorders (STD)" Subscale Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Sleep Disorders Scale for Children (SDSC) is a 26-item, parent-reported measure used to screen for sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Sleep-Wake Transition Disorders (STD) Subscale (items 6, 7, 8, 12, 18, and 19). The sum of the 6 items yields the raw Subscale score (range: 6 to 30; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 46
score on a scale | -0.3 (2.64)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.4385, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

24. Secondary Outcome: Change From Baseline in Sleep Disorders Scale for Children (SDSC) "Disorders of Excessive Somnolence" (DES) Subscale Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency: 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Disorders of Excessive Somnolence (DES) Subscale (items 22, 23, 24, 25, and 26). The sum of the 5 items yields the raw Subscale score (range: 5 to 25; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 46
score on a scale | 0.4 (3.75)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.5073, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

25. Secondary Outcome: Change From Baseline in the Sleep Disorders Scale for Children (SDSC) "Sleep Hyperhidrosis (SH)" Subscale Scores at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Sleep Disturbance Scale for Children (SDSC) is a 26-item, parent-rated scale that assesses the presence of sleep disturbances in children/adolescents. All items are rated on a 5-point scale based on past week; Item 1, average sleep duration: 1 = "9-11 h" to 5 = "less than 5 h"; Item 2, average sleep latency, 1 = "less than 15 min" to 5 = "more than 60 min"); Items 3-26, sleep disturbances: 1 = "Never" to 5 = "Always". Six subscale scores are generated, including the Sleep Hyperhidrosis (SH) Subscale (items 9 and 16). The sum of the 2 items yields the raw Subscale score (range: 2 to 10; the higher the score, the more severe the disturbance). Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 46
score on a scale | 0.0 (1.32)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.9119, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

26. Secondary Outcome: Change From Baseline in Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) Total Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) is a validated, 11-item scale for the assessment of ADHD-related morning and evening behaviors impacting at-home functioning in children with ADHD. There are 3 items related to morning behaviors and 8 items related to evening behaviors. The parent/guardian rates each item on a 4-point scale based on their child's behavior during the past week, where 0 = "no difficulty" to 3 = "a lot of difficulty". The sum of all 11 items yields a Total score (range: 0-33); the higher the score, the more severe the impairment/difficulty. Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: Safety population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data is summarized by number of subjects analyzed (n; subjects with a valid Weekly Parent Rating of Evening and Morning Behavior-Revised [WPREMB-R] assessment at baseline [pre-dosing], Week 4, and Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 47
score on a scale | -2.4 (6.40)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.0140, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

27. Secondary Outcome: Change From Baseline in Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) "Morning Behaviors" Subscale Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) is a validated, 11-item scale for the assessment of ADHD-related morning and evening behaviors impacting at-home functioning in children with ADHD. There are 3 items related to morning behaviors and 8 items related to evening behaviors. The parent/guardian rates each item on a 4-point scale based on their child's behavior during the past week, where 0 = "no difficulty" to 3 = "a lot of difficulty". The sum of all 3 items related to morning behaviors yields a WPREMB-R Morning Behaviors Subscale score (range: 0-9); the higher the score, the more severe the impairment/difficulty. Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 47
score on a scale | -0.5 (2.22)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.1542, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

28. Secondary Outcome: Change From Baseline in Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) "Evening Behaviors" Subscale Score at Week 4 (AM Dosing) Versus at Week 8 (PM Dosing)
Description: The Weekly Parent Rating of Evening and Morning Behavior-Revised (WPREMB-R) is a validated, 11-item scale for the assessment of ADHD-related morning and evening behaviors impacting at-home functioning in children with ADHD. There are 3 items related to morning behaviors and 8 items related to evening behaviors. The parent/guardian rates each item on a 4-point scale based on their child's behavior during the past week, where 0 = "no difficulty" to 3 = "a lot of difficulty". The sum of all 8 items related to evening behaviors yields a WPREMB-R Evening Behaviors Subscale score (range: 0-24); the higher the score, the more severe the impairment/difficulty. Raw score is converted to a change from baseline (CFB) score. A mean difference (the Week 8 minus the Week 4 CFB score) <0 represents a better outcome at Week 8.
Time Frame: Week 4 and Week 8
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 47
score on a scale | -1.9 (4.78)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4 versus Week 8; Test type: Other; p = 0.0086, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

29. Secondary Outcome: Change From Baseline in the "Morning" Parent-rated ADHD Rating Scale, 5th Edition (PR-ADHD-RS-5) Total Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Parent/guardian rates each item on a 4-point scale from 0 (never or rarely) to 3 (very often) based on observations of their child's behavior during the morning hours in the past week. The raw Total score (sum of 18 items range: 0-54; the higher the score, the more severe the ADHD symptoms in morning hours), is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data at each Week/Visit is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid "Morning" Parent-rated ADHD Rating Scale, 5th Edition [PR-ADHD-RS-5] assessment at baseline [pre-dosing] and at Week 4 or Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 50
  Raw score; Baseline | 32.6 (12.10)
  Change from Baseline score; Week 4: number analyzed (Participants) | 39
  Change from Baseline score; Week 4 | -10.2 (11.90)
  Change from Baseline score; Week 8: number analyzed (Participants) | 37
  Change from Baseline score; Week 8 | -12.0 (14.28)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

30. Secondary Outcome: Change From Baseline in "Evening" Parent-rated ADHD Rating Scale, 5th Edition (PR-ADHD-RS-5) Total Score at Week 4 (AM Dosing) and at Week 8 (PM Dosing)
Description: The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Parent/guardian rates each item on a 4-point scale from 0 (never or rarely) to 3 (very often) based on observations of their child's behavior during the evening hours in the past week. The raw Total score (sum of 18 items range: 0-54; the higher the score, the more severe the ADHD symptoms in morning hours), is converted to a change from baseline (CFB) score. A CFB score <0 represents a better outcome.
Time Frame: Baseline, Week 4, and Week 8
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data at each Week/Visit is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid "Evening" Parent-rated ADHD Rating Scale, 5th Edition [PR-ADHD-RS-5] assessment at baseline [pre-dosing] and at Week 4 or Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 56
score on a scale
  Raw score; Baseline: number analyzed (Participants) | 47
  Raw score; Baseline | 33.6 (10.50)
  Change from Baseline score; Week 4: number analyzed (Participants) | 37
  Change from Baseline score; Week 4 | -9.6 (11.24)
  Change from Baseline score; Week 8: number analyzed (Participants) | 26
  Change from Baseline score; Week 8 | -14.3 (11.62)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Open-Label Treatment; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

31. Secondary Outcome: Change in Baseline in the "Morning" Versus "Evening" Parent-rated ADHD Rating Scale, 5th Edition (PR-ADHD-RS-5) Total Score at Week 4 (AM Dosing)
Description: The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Parent/guardian rates each of 18 items on the "Morning" PR-ADHD-RS-5 and each of 18 items on the "Evening" PR-ADHD-RS-5 on a 4-point scale from 0 (never or rarely) to 3 (very often) based on observations of their child's behavior during the morning hours in past week and evening hours in the past week, respectively. For each assessment, the raw Total score (sum of 18 items; range: 0-54; the higher the score, the more severe the morning or evening ADHD symptoms) is converted to a change from baseline (CFB) score. A mean difference (the Evening minus the Morning CFB score) <0 represents a better outcome in the Evening.
Time Frame: Week 4
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data is summarized with by number of subjects analyzed (n; subjects with a valid "Morning" and "Evening" Parent-rated ADHD Rating Scale, 5th Edition [PR-ADHD-RS-5] assessment at baseline [pre-dosing] and Week 4). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 33
score on a scale | 1.1 (10.59)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 4; "Morning" PR-ADHD-RS-5 Total score versus "Evening" PR-ADHD-RS-5 Total score; Test type: Other; p = 0.5582, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

32. Secondary Outcome: Change in Baseline in the "Morning" Versus "Evening" Parent-rated ADHD Rating Scale, 5th Edition (PR-ADHD-RS-5) Total Score at Week 8 (PM Dosing)
Description: The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Parent/guardian rates each of 18 items on the "Morning" PR-ADHD-RS-5 and each of 18 items on the "Evening" PR-ADHD-RS-5 on a 4-point scale from 0 (never or rarely) to 3 (very often) based on observations of their child's behavior during the morning hours in past week and evening hours in the past week, respectively. For each assessment, the raw Total score (sum of 18 items range: 0-54; the higher the score, the more severe the morning or evening ADHD symptoms) is converted to a change from baseline (CFB) score. A mean difference (the Evening minus the Morning CFB score) <0 represents a better outcome in the Evening.
Time Frame: Week 8
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least one dose of SPN-812. Data is summarized by number of subjects analyzed (n; subjects with a valid "Morning" and "Evening" Parent-rated ADHD Rating Scale, 5th Edition [PR-ADHD-RS-5] assessment at baseline [pre-dosing] and Week 8). Due to attrition and/or missing data, the number of subjects analyzed may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 23
score on a scale | -1.6 (11.41)
Statistical Analysis 1: Comparison: Open-Label Treatment; Week 8; "Morning" PR-ADHD-RS-5 Total score versus "Evening" PR-ADHD-RS-5 Total score; Test type: Other; p = 0.5061, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) were collected after the first dose administration at Baseline visit up to nine weeks (i.e., safety follow up phone call 1 week after end of study visit).
Description: Treatment Emergent Adverse Event (TEAE) is an adverse event (AE) with a start date on or after the first dose of study medication is taken, or that worsened following first administration of study medication. Since the same subjects progress through Weeks 1 - 8, the same subject may be counted in Week 1 - 4, Week 5 - 8, Overall Duration, and Post treatment.
Groups:
- Open-Label Treatment: Subjects 6-11 years of age: 100 to 400mg SPN-812 (100 mg oral capsule)
  Subjects 12-17 years of age: 100 to 600mg SPN-812 (100 mg, 200 mg oral capsule)
  SPN-812: Viloxazine extended-release capsule
Arm/Group | Open-Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 32/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Treatment (N=56)
Headache (Nervous system disorders) | 10 (10)
Decreased Appetite (Metabolism and nutrition disorders) | 7 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6)
Insomnia (Nervous system disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Irritability (Psychiatric disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04786990/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT04786990/SAP_003.pdf